CLINICAL TRIAL: NCT05527587
Title: Examining the Effects of an 8-Week Open Label Nature-Based Park Visit Program on the Quality of Life, Behaviors and Cognitive Symptoms of Individuals With Dementia and Their Caregivers
Brief Title: The Effects of a Park Visit Program on Individuals With Dementia and Their Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB22-0788
Record Dates: First submitted 2022-08-22; First posted 2022-09-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-08

CONDITIONS: Mild Dementia; Moderate Dementia; Alzheimer Disease
Keywords: Dementia; Nature; Outdoor activities; Mental health; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychological Well-Being

STUDY DESIGN:
Masking Description: Since we have limited evidence on the effects of non-pharmacological treatment for dementia including nature-based activities, we would like to perform an open-label pilot study to understand the effects of nature-based activities in people living with dementia in preparation for a future controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nature Connections Group (Experimental): Participants will be screened to confirm their eligibility to partake in the study. Participants who meet the study criteria will then be invited to participate in the nature connections intervention. At the start of the intervention, mid-intervention and post intervention, participants will be invited to participate in assessments of their behaviour and mood symptoms, cognition, quality of life, caregiver burden and stress levels using different measures and questionnaires at the University of Calgary. Participants will be provided with a visit passport to record a log of activities completed during the park visits.
  Interventions: Other: Nature Connections Intervention

INTERVENTIONS:
Other: Nature Connections Intervention — 10 PLWD and their 10 caregivers will be examined for the effects of a park visit program on their behaviour and mood symptoms, cognition, and quality of life over the period of 8-weeks. If participants meet the study criteria, an initial education session on the health benefits of nature will be provided to the them. Participants will then be invited to participate in the park visit program which will have them visiting local parks or outdoors spaces with their caregivers. They will be encouraged to allocate approximately 120 minutes each week to outdoor park activities for 8 weeks. Participants will be provided with a visit passport to record a log of activities completed during the park visits. During the 8 weeks of intervention, participants will also participate in a weekly check-in meeting with other participants to discuss about their experiences with the park visits.
  Other Names: Park Visit Program; Nature-based Activities

SUMMARY:
The overall goals of our project is to understand the effects of participating in park visits and nature-based activities for people living with dementia and their caregivers. Nature-based activities such as park visits can have beneficial effects on quality of life, psychological symptoms and physical health. However, there may be barriers for people with dementia and their caregivers that may prevent them from engaging in park visits. The Nature Connections park visit program will provide education sessions for 10 persons living with dementia and 10 caregivers highlighting the beneficial effects of park visits and address common barriers to participating in park visits. Following the education session participants will be provided with weekly telephone/internet support meetings for participants to share their experiences with park visits and to address any challenges individuals encountered when trying to complete their visits. The impact of park visits on quality of life, behaviours, and measures of stress for people with dementia and their caregivers will be assessed over 8 weeks. Following completion of the program participants will provide an evaluation of the program to understand their experience and satisfaction with the program. This project will provide new information about the effects of park visits as a practical strategy to improve the quality of life, psychological symptoms and measures of stress for both people with dementia and caregivers.

DETAILED DESCRIPTION:
Background & Rationale:

Cognitive impairment has been the main focus in treating and caring for people living with dementia (PLWD). More recently, non-cognitive symptoms associated with dementia are increasing and forcing families to seek non-pharmacological treatment approaches for dementia related symptoms. Previous studies has also shown the effect of aerobic exercises and other non-pharmacological interventions in providing a range of benefit such as physical, mental, and emotional benefit in people without dementia, however, there is limited evidence on the effect of nature-based activities on PLWD. Many PLWD are disconnected from the outdoors due to a significant amount of time spent indoors resulting in reduced knowledge about how nature-based activities can benefit the QoL of PLWD. The specific aim of this project is to evaluate the effect of parks visit, an example of nature-based activities on the neuropsychiatric symptoms, QoL, cognition, stress and burden of PLWD and their caregivers.

Objectives:

1) The objective of this project is to investigate the impact of a 8-week nature park visit program intervention on stress, quality of life and cognition in 10 pairs of PLWD and their caregivers; 2) Evaluate the impact of potential barriers on participation in activity and their influence on the QoL of PLWD.

Methods:

10 pairs of PLWD and their caregivers who live in the community will be recruited into the nature connections intervention program. This study will be an open-label pilot study using pre-post design. The nature connections intervention will include an 8-week park visit program after which PLWD and their caregivers will be assessed on factors including changes in cognitive function, changes in mood and behaviors, changes in QoL, and changes in stress levels. These factors will be assessed in participants at baseline, week 4 (mid-intervention) and week 8 (post-intervention) to appropriately evaluate the impact of the intervention. Screening measures including demographics, cognition, physical activity, and functional ability will be assessed and collected during the screening period to meet the inclusion criteria for the study. Behavior and mood symptoms will be assessed using the Neuropsychiatric Inventory-Questionnaire (NPI-Q while depressive symptoms will be assessed using the Cornell Scale for Depression in Dementia (CSDD). Cognition will be measured using the Repeatable Battery for Assessment of Neuropsychological Syndromes (RBANS). Changes in Quality of life will be assessed using the Dementia Quality of Life (DEMQOL) assessment. The activity log of park visits will be recorded from baseline until week 8. Caregiver specific outcomes, caregiver burden and caregiver well-being and support will be assessed at baseline, week 4 during intervention and week 8 post intervention. Caregiver burden will be assessed using the Zarit Burden Interview (ZBI) while caregiver well-being and support will be measured using the Carer Well-being and Support questionnaire. The intervention will also include weekly check-in meetings where participants can discuss their experience with the park visits with other participants.

Data Analysis:

The primary outcome for PLWD is change in neuropsychiatric symptoms as measured from baseline to week week 8 on the NPI-Q using paired t-tests. Secondary outcomes include measurement of depressive symptoms (CSDD), cognition (RBANS), quality of life, care giver stress and caregiver burden (ZBI) at weeks 4 and week 8 of the study. Two-sided p-values of <0.05 will be used as the threshold for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are 65 years or older
* PLWD who meet Diagnostics and Statistical Manual of Mental Disorders DSM-5 for major neurocognitive disorder due to Alzheimer's disease
* Individuals with mild to moderate dementia as assessed on the Montreal Cognitive Assessment (MoCA) corresponding to scores of 12-25 on the 12-item assessment or 10-18 on the 9-item telephone MoCA assessment
* Participants who currently participate in less than 2 hours of outdoor activities weekly using the Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire
* Caregivers who spend at least 2 hours per week with PLWD
* Participants that are able to mobilize independently or with assistive devices and have the ability access local parks either independently or with the assistance of caregivers.

Exclusion Criteria:

* Participants with unstable conditions that prevent outdoor activities
* Patients residing in long-term care or nursing homes
* Individuals with AD who have no access to a caregiver
* Participants with limited mobility that prevents outdoor activities
* Participants who do not have adequate comprehension and verbal communication in English necessary to participate in measurement of outcomes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Symptoms | Change from Baseline Neuropsychiatric Symptoms at 8 weeks (post-intervention)
  The primary measure of neuropsychiatric symptoms is mood and behavior measured at week 8 as measured on the Neuropsychiatric Inventory Questionnaire (NPI-Q) total score. This questionnaire measures severity of the symptoms in individuals on a 3-point scale (1=mild; 2=moderate; and 3=severe) and the distress associated with the symptoms on a 5-point scale (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=extreme distress). The scores range from 0 (absence of behavioral symptoms) to 144 points (maximum severity of behavioral symptoms)

SECONDARY OUTCOMES:
Depressive Symptoms | Change from Baseline Depressive symptoms at 4 weeks (mid-intervention) and at 8 weeks (post-intervention)
  Depressive symptoms which will be measured using Cornell Scale for Depression in Dementia. This scale assesses signs and symptoms of major depression in PLWD via a caregiver reported proxy. There are 19 items on the scale, each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 are associated with absence of significant depressive symptoms. The CSDD total score will be used to assess change in depressive symptoms.
Cognition | Change from Baseline Cognition at 4 weeks (mid-intervention) and at 8 weeks (post-intervention)
  Cognition which will be measured using the Repeatable Battery for Assessment of Neuropsychological Syndromes (RBANS). This is a brief, individually administered test to measure the rate of cognitive decline or improvement. This assessment consists of 12 subtests, which yield five Index scores and a total Scale score. The scores are classified based on the following: average/mild impairment (standard scores of 70 or above), moderate impairment (standard scores from 55 to 69), and severe impairment (standard scores <54)). The RBANS total score will be used to measure change in cognition.
Quality of Life assessed by DEMQoL (Dementia Quality of Life assessment) | Change from Baseline Health-related quality of life at 4 weeks (mid-intervention) and at 8 weeks (post-intervention)
  Quality of life will be assessed using the dementia quality of life assessment.These are interviewer-administered measures which obtain self- and caregiver reports of the health-related quality of life for people with dementia. Items inquire about 'feelings', 'memory' and 'everyday life' of the person with dementia in the last week. Each question is assessed on a 4-point scale (a lot, quite a bit, a little, not at all). The items are scored according to a standard scoring to produce an overall score where higher scores represent better health-related quality of life. The DEMQoL total score ranges from 28 to 112.
Caregiver Burden | Change from Baseline Caregiver Burden at 4 weeks (mid-intervention) and at 8 weeks (post-intervention)
  Caregiver burden will be assessed using the Zarit Burden Interview scale. This consists of 22 items, each item on the interview is a statement which the caregiver is asked to endorse using a 5-point Likert scale (0=never, 1=rarely, 2=sometimes, 3=quite frequently, 4=nearly always). The sum of scores range between 0-88 (0 - 21 little or no burden; 21 - 40 mild to moderate burden; 41 - 60 moderate to severe burden; 61 - 88 severe burden).
Caregiver Well-being and Support | Change from Baseline Caregiver well-being and support at 4 weeks (mid-intervention) and at 8 weeks (post-intervention)
  Caregiver well-being and support will be measured using the carer well-being and support questionnaire. This questionnaire contains two subscales: wellbeing and support. Higher well-being scale total (range: 0-128) indicates better carer wellbeing; while higher support scores (reverse scoring used and total range: 0-51) indicates lower satisfaction with support received.
Neuropsychiatric Symptoms | Change from Baseline to week 4 on the NPI-Q total score.
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) measured at week 4 will be included as a secondary outcome and the NPI-Q properties are described in the primary outcome section of the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Dallas P Seitz, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Cumming School of Medicine, University of Calgary, Calgary, Alberta, Canada